CLINICAL TRIAL: NCT06527924
Title: A Randomized Controlled Trial of the Difference in Sagittal Angle of the Lower Limbs Between Healthy Individuals and Patients With Osteoarthritis
Brief Title: A Randomized Study on Sagittal Angle Differences in Lower Limbs Between Normal Individuals and Osteoarthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Jiafeng Yi, Resident doctor, Chinese PLA General Hospital
Other Study IDs: 2023KY024-KS001
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: OA; TKA; EOS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health Group: Non-osteoarthritis (OA) patients who underwent sagittal plane EOS examinations at the Chinese PLA General Hospital between September 2024 and September 2026.
- OA group: OA patients who underwent sagittal plane EOS examinations at the Chinese PLA General Hospital from September 2024 to September 2026. The sagittal alignment angles on the EOS radiographs of the subjects were measured to establish a classification system for extension or non-extension.

SUMMARY:
With China gradually entering an aging society, the proportion of the elderly population is gradually increasing, and the number of patients with knee disease is also increasing year by year. Total knee arthroplasty is one of the effective methods for the treatment of joint disease, which can effectively relieve knee pain, restore function and improve the quality of life. The goal of total knee arthroplasty is to relieve pain, restore function and obtain a long service life. Whether total knee arthroplasty can obtain good alignment is very important for the postoperative recovery of patients. The alignment of lower limb sagittal position is of great significance for evaluating whether the crowd is straightened or not, and can also evaluate and guide the TKA in sagittal position. At present, there are few studies on the sagittal position of the lower limb, and there is no clear definition of whether the lower limb is extended in the sagittal position. At the same time, there is no clear method to evaluate whether the lower limb is extended in the sagittal position in normal people and patients with OA. Therefore, it is urgent to develop a classification standard for the sagittal extension of the lower limb, which can be used in clinical evaluation and TKA operation evaluation. This study will be carried out in the first medical center of the Chinese PLA General Hospital, and a total of about 400 people are expected to be enrolled.

DETAILED DESCRIPTION:
I. Clinical Research Background As China enters an aging society, the elderly population is increasing, leading to a rise in knee joint disease patients. Total knee arthroplasty is an effective treatment for joint disorders, alleviating knee pain, restoring function, and improving quality of life.The objectives of total knee arthroplasty are to relieve pain, restore function, and ensure a long-lasting implant. Achieving good alignment is crucial for patient recovery after total knee arthroplasty. The alignment of the lower limb in the sagittal plane is important for assessing whether the limb is extended or not, which also guides the sagittal alignment during TKA. Currently, there is limited research on the sagittal alignment of the lower limb, and there is no clear definition of whether the lower limb should be extended in this plane. Additionally, existing studies lack a clear method for assessing sagittal alignment in both normal individuals and patients with OA. Consequently, there is an urgent need to establish a classification standard for sagittal alignment of the lower limb, applicable to clinical and TKA surgical evaluations.

II. Content of Clinical Trials (I) Overall Design and Sample Size This study is a prospective clinical investigation, encompassing two groups: ① Healthy Group: Non-osteoarthritis (OA) patients who underwent sagittal plane EOS examinations at the People's Liberation Army General Hospital between September 2024 and September 2026. ② OA Group: OA patients who underwent sagittal plane EOS examinations at the same hospital from September 2024 to September 2026. The sagittal alignment angles on the EOS radiographs of the subjects were measured to establish a classification system for extension or non-extension.

(II) Randomization and Control in the Study Randomized controlled trial. (III) Content From September 2024 to September 2026, at the Chinese PLA General Hospital, a cohort of 200 non-lower limb-related non-osteoarthritis (OA) patients who underwent sagittal plane EOS imaging was studied. Basic demographic data, including age, weight, and height, were recorded. An experienced researcher measured angles such as the modified mechanical axis angle, femoral anterior bowing angle, and tibial plateau posterior slope angle. The collected data underwent statistical analysis to determine the 95% normal distribution ranges for these angles, thereby establishing the sagittal plane ranges for 'extension,' 'overextension,' and 'extension-limited' in the knee joint. Additionally, 200 OA patients attending the director's outpatient clinic were measured by the researcher and taken to the radiology department for sagittal plane imaging according to the established EOS requirements. The same three angles were measured and recorded, and the aforementioned classification was used to assess whether the OA patients were in extension or not. The differences between the two groups were then compared.

III: Trial Procedure (I) Subject Enrollment Physicians selected subjects who underwent EOS imaging at our hospital from September 2024 to September 2026, and screened them based on inclusion and exclusion criteria. If a patient met the inclusion criteria, the details of the research project were thoroughly explained to them, and they were required to sign the relevant informed consent form.

(II) Methodology Subjects who met the inclusion criteria and underwent sagittal EOS examinations at the Radiology Department of the First Medical Center of the Chinese PLA General Hospital from September 2024 to September 2026 were included in the study. Imaging data were collected under the following conditions: ① the radiographer stood on one leg; ② the two femoral condyles coincided on the lateral radiograph. Basic demographic information, including age, weight, and height, was recorded. An experienced researcher measured angles such as the modified mechanical axis angle, femoral anterior bowing angle, and tibial plateau posterior slope angle. The obtained data were subjected to statistical analysis to determine the 95% normal distribution range values for these three angles, thereby establishing the angular ranges for "extension," "hyperextension," and "limited extension" of the knee joint in the sagittal plane. A total of 200 OA patients attending the outpatient clinic of director were measured by the researcher, who then brought them to the radiology department to undergo sagittal radiography according to the established EOS imaging requirements. The same three angles were measured and recorded, and the aforementioned classification was used to evaluate whether the OA patients were in extension or not. The differences between the two groups were compared.

(III) Clinical Evaluation Indices

(1) Primary Observational Indicators:

1. Sagittal plane femur lateral, tibia lateral modified mechanical axis angle; angle formed by the line connecting the center of the femoral head, the center of the ankle joint, and the hinge point of the knee joint;
2. Sagittal plane femoral anterior arch angle;
3. Sagittal posterior slope angle of the tibial plateau;
4. Coronal Hip-Knee-Ankle Angle (HKA), Lateral Distal Femoral Angle (LDFA), Medial Proximal Tibial Angle (MPTA).

(2) Secondary Observational Indicators

1) Basic demographic profile of the patient. (IV) Case Report Documentation Researchers should diligently complete all research documentation, including the verification of all participants (capable of effectively collating diverse record-keeping materials, such as case report forms and original hospital records), all original signed patient informed consent forms, and detailed records of all case report forms. Upon the conclusion of the trial, all clinical research materials shall be transferred to the Clinical Research Organization's office for safekeeping.

Ⅳ: Statistical Analysis Methods All results were computed using SPSS 26.0. A comprehensive listing of all collected data will be presented, followed by a descriptive summary of the data. Categorical variables will be summarized using frequencies and percentages, while continuous variables will be summarized by the number of subjects, mean, mean difference relative to baseline (if applicable), median, standard deviation, 95% confidence intervals, minimum, and maximum values at each assessment time point.

Prior to database lock, the definitive statistical analysis plan will be established, and the pertinent clinical and statistical personnel will document their decisions regarding the inclusion or exclusion of data from each subject.

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 80 years old;
2. Non OA examinees of lower limb sagittal EOS in the General Hospital of Chinese PLA;
3. OA patients with sagittal EOS were photographed in the Department of joint surgery, General Hospital of Chinese PLA;
4. Patients are willing to participate in the study and sign written informed consent.

Exclusion Criteria:

1. People unable to conduct EOS inspection;
2. Combined with knee meniscus injury, anterior cruciate ligament injury and other diseases that may affect the sagittal force line of the knee joint
3. Combined with other diseases that may affect the study
4. Patients refused to use their imaging data and knee score for this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non OA patients and OA patients undergoing EOS in our hospital from September 2024 to September 2026.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Sagittal plane femur lateral, tibia lateral modified mechanical axis angle. | From admission to discharge, up to 1 week
Angle formed by the line connecting the center of the femoral head, the center of the ankle joint, and the hinge point of the knee joint. | From admission to discharge, up to 1 week
Sagittal plane femoral anterior arch angle. | From admission to discharge, up to 1 week
Sagittal posterior slope angle of the tibial plateau. | From admission to discharge, up to 1 week
Coronal Hip-Knee-Ankle Angle (HKA) | From admission to discharge, up to 1 week
Lateral Distal Femoral Angle (LDFA) | From admission to discharge, up to 1 week
Medial Proximal Tibial Angle (MPTA) | From admission to discharge, up to 1 week

SECONDARY OUTCOMES:
Basic demographic profile of the patient | From admission to discharge, up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chai, doctorate, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China